CLINICAL TRIAL: NCT04414527
Title: Effects of Video-based Health Education on Health Status of Pregnant Mothers and Their Infants (From 0 to 6 Months) in Dirashe District Southern Ethiopia - a Cluster Randomized Controlled Trial.
Brief Title: Effects of Video-based Health Education on Maternal and Child Health in Ethiopia
Acronym: MCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Flemish Interuniversity Council (VLIR) (Network); Arba Minch University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BC-06756
Record Dates: First submitted 2020-04-21; First posted 2020-06-04 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Anemia; Antenatal Care; Birth Outcomes; Worm Infection; Bacterial Vaginoses; Exclusive Breastfeeding
Keywords: Video-based behavior change communication; Iron and folic acid supplementation; Antenatal care; Soil transmitted helminths; Bacterial vaginoses; Exclusive breastfeeding
MeSH Terms: conditions — Anemia; Trematode Infections; Vaginosis, Bacterial; Breast Feeding

STUDY DESIGN:
Intervention Model Description: In a two-arm cluster randomized trial, 675 eligible pregnant women in their first trimester (12 weeks of gestation) will be recruited and followed up until delivery, and in pair with their infant up-to six months postpartum.
  1. Eligible pregnant women in the intervention group will receive video-based nutritional and hygienic education package (Health-Video) for six months until delivery and then for another six-month postpartum.
  2. Pregnant women in the control group will receive the standard education package as per the Ethiopian guidelines.
  The intervention will include home-to-home visit for delivery of healthy nutrition and hygiene messages using prepared video-based messages, and participation in monthly forums facilitated by nurses using also videos for demonstration of nutritional and hygienic care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard counseling (Other): Pregnant women in the control group will receive the standard education package as per the Ethiopian guidelines. In the standard health care, pregnant women receive a minimum of four ante-natal care visits at the health centers during which they also receive iron and folic acid supplementation. They participate in monthly forums facilitated by nurses to answer questions and concerns regarding nutritional care.
  Interventions: Behavioral: Standard counselling
- Health-Video (Experimental): Women in the Health-Video group will receive home visits for delivery of healthy nutrition messages using prepared video-based messages every two weeks. They will also participate in monthly forums facilitated by nurses using also videos for demonstration of nutritional care. During the monthly forums (six in total during the pregnancy and the post-partum periods), the messages will all be given as a video show coordinated by a nurse/ health professional for any questions. During postnatal period, two counseling sessions will be delivered within two weeks of birth, and 12 sessions or twice every month till 6 months.
  Interventions: Behavioral: Health-Video

INTERVENTIONS:
Behavioral: Standard counselling — The control cohort will receive national standard counseling during four ante-natal care visits.
  Women in the control group will receive additionally
  1. national nutrition and health care including IFA supplementation,
  2. treatment of any symptomatic health condition and deworming in case of symptomatic complaints during second and third trimesters,
  3. Women who experience odor, itching or discharge will be treated for candidiasis and bacterial vaginosis.
  Other Names: Control
  Arms: Standard counseling
Behavioral: Health-Video — The intervention cohort Health-Video will receive innovative video-based nutritional and hygienic education.
  Women in this group will receive additionally:
  1. National nutrition and health care including IFA supplementation
  2. treatment of any symptomatic health condition and deworming in case of symptomatic complaints during second and third trimesters,
  3. Women who experience odor, itching or discharge will be treated for candidiasis and bacterial vaginosis.
  Other Names: Video-based counselling
  Arms: Health-Video

SUMMARY:
Low adherence to recommended health and nutrition strategies during the critical 1000 day-window of opportunity is multifactorial but low quality communication is key limitation. Innovative strategies to improve interpersonal communication can reduce the burden and the fatigue of community health workers and may result in a greater change. The findings of this project will support governments and other stakeholders in their delivery of high impact nutrition and health practices.

This intervention aims to improve adherence to ante- and post-natal care practices and recommendations by the use of our video-based health education. These videos will be implemented through home-based counseling by trained assistants, and video-based forum participation led by community nurses and health extension workers (HEWs). During the monthly forums, the educational package will be delivered in a video form - locally prepared using multiple approaches like testimony, comedy, dramas in the form of questions and answers, group discussions and deductive approaches. Cordless projectors and locally created videos give the health community more quality control over the end message, expand the number of people reached, allow for the use of minimally trained non-expert facilitators such as the hews, and allow for contextually appropriate information. They can also be used in areas without access to electricity, helping to bridge the digital divide, and serving as a leapfrog technology for areas that would otherwise not have access to media.

DETAILED DESCRIPTION:
In Ante- and post-natal care, low adherence to recommended health and nutrition strategies during the critical 1,000 day-window of opportunity is multifactorial, but low-quality communication is key limitation. Innovative strategies to improve interpersonal communication can reduce the burden and the fatigue of community health workers and may result in a greater change. The findings of this project will support governments and other stakeholders in their delivery of high impact nutrition and health practices.

Focused antenatal care (FANC), including iron and folic acid supplementation (IFA) is one of the main strategies to reduce maternal and child deaths. The WHO recommends at least four hospital visits during the pregnancy. Supplementation with IFA during pregnancy improves birth weight and reduces megaloblastic anemia by 79%. The uptake of nutritional and health practices is influenced by complex, contextual determinants at the individual and community levels. Evidence showed that Social and Behavior Change Communication (SBCC) is an effective approach to increase the uptake of key strategies and to sustain behavior change.

Ethiopia, a low-income country in sub-Saharan Africa, has one of the highest maternal and infant mortality rates. It is estimated that 676 mothers die per 100,000 live births and that 59 infants die per 1,000 live births. Maternal anemia is associated with an increased risk of maternal death. Iron deficiency anemia is a strong risk factor for low birthweight (LBW) and perinatal mortality. genital infections such as bacterial vaginosis, candidiasis and worm infections (such as intestinal hookworm infections) are considered important infections that possibly could confound the study results. Bacterial vaginosis and candidiasis are a known risk factor for preterm birth. these infections are also linked with anemia and maternal nutritional status. Hookworm infections are highly prevalent in Ethiopia and are associated with undernutrition and anemia.

The reports of the Ethiopian Demographic and Health Survey showed an increase in women aged 15-49 years in Ethiopia receiving antenatal care (ANC) from a skilled provider up to 62% in 2016 (EDHS, 2016). The percentage of women taking IFA supplements for 90 days or more remains at a substandard level of only 5% (EDHS, 2016). Antenatal care coverage for at least one visit is 28% but coverage for at least four visits declines to 12%, suggesting systemic barriers that potentially prevent the mothers from returning to the health centers. One of the barriers may be perceived failure of the existing interventions to make a meaningful impact that could stimulate the desired behavioral change.

This intervention aims to improve adherence to ante- and post-natal care practices and recommendations by the use of our video-based health education. These videos will be implemented through home-based counseling by trained assistants, and video-based forum participation led by community nurses and Health Extension Workers (HEWs). The nutrition-specific education packages will be based on the WHO-UNICEF key messages booklet on the community, infant and young child feeding counseling package and will be culturally adjusted to fit the local context and translated into the main four local languages. The videos will also include some hygienic aspects that reduce the risk of both genital and parasitic infections, that are also causing undernutrition, anemia and/or adverse pregnancy outcomes. During the monthly forums, the educational package will be delivered in a video form - locally prepared using multiple approaches like testimony, comedy, dramas in the form of questions and answers, group discussions and deductive approaches (more details can be found on OMPT website https://www.ompt.org/).

The main objective of this project is to assess the effects of this innovative video-based health education on reproductive health, and on birth outcomes and the nutritional status of women and their infants from birth to six months of age.

PRIMARY OBJECTIVES

1. To assess the effects of video-based health education package provided to pregnant and lactating women on the knowledge, attitude and practice on recommended health including adherence to ANC visits and to IFA supplementation.
2. To assess the effects of video-based health education on birth outcomes and anemia status of women during pregnancy, at delivery and six-month postpartum.
3. To evaluate the effect of video-based health education on early initiation and exclusive breastfeeding (EBF) of infants from 0-6 months of age In this two-arm cluster randomized trial, 675 pregnant women in their first trimester (12 weeks of gestation) will be recruited and followed up until delivery and then with their infants for six months postpartum.

The intervention will include home to home visit for delivery of healthy nutrition and hygienic messages using prepared video-based messages. participation in monthly forums will be facilitated by nurses using also videos for demonstration of nutritional and hygienic care and will be delivered at the homes of the participants every month by trained HEW until delivery, in addition to the ANC regular visits. During the monthly forums (six in total during the pregnancy and the post-partum periods), the messages will all be given as a video show, coordinated by a nurse/ health professional who will further answer any questions. During the postnatal period, two counseling sessions will be organized within the first two weeks after birth, and a further six sessions ( every month) till 6 months postnatally.

The HEW will distribute the IFA 30 tablets (30 mg elemental iron and 400 µg of folic acid) every month, and will provide counseling on the importance of- and instructions on adherence and other recommendations as detailed earlier. Pregnant women in the control group will receive the standard education package as per the Ethiopian guidelines. In the standard health care, pregnant women receive a minimum of four ANC visits at the health centers during which they also receive IFA supplementation. The control and the intervention groups receive the same amount of tablets (i.e. 30 tablets containing 30 mg elemental iron and 400 µg of folic acid, every month). Monthly IFA utilization will be checked through HEW or our trained service delivery workers during home to home visit. Women who test positive for soil-transmitted helminth will be treated according to the national protocol starting from the second trimester (treatment is not advised during the first trimester). Women who experience odor, itching or discharge will be treated for candidiasis and bacterial vaginosis.

Data will be collected in pregnant women at baseline, at six and at 9 months of pregnancy . After delivery data will be collected in the pairs mother-infant within two weeks and at 3 and 6 months postpartum. At the different time points, biological samples will be collected to assess the micronutrient status, the presence of inflammations and the presence of genital and parasitic infections.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Aged at least 18 years
* Permanent resident of the village of the study intervention/control
* Planned availability during the whole period of the study (12 months)
* Acceptance of the intervention package including home visits for data collection and morbidity follow up.

Exclusion Criteria:

* Severe anemia (hemoglobin <70 g/L),
* Under nutrition (defined as body mass index before pregnancy of <18.5 kg/m2),
* Chronically ill mothers with tuberculosis or other chronic diseases,
* Reported HIV-positive mother.
* Individuals with anatomical deformity will be excluded due to the difficulty of measurement of height.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Adherence to iron and folic acid supplementation during pregnancy | Monthly during six months pregnancy
  Monthly disappearance rate of IFA tablets
Adherence to iron and folic acid supplementation post-partum | Monthly during three months postpartum
  Monthly disappearance rate of IFA tablets
Maternal anemia during pregnancy | Hemoglobin concentrations will be measured at 9 months pregnancy
  Hemoglobin concentrations (g/dL)
Maternal anemia post-partum | Hemoglobin concentrations will be measured at six months postpartum
  Hemoglobin concentrations (g/dL)
Early initiation | At birth (six months after the enrollment)
  Prevalence of newborns put to the breast in the first hour after birth
Exclusive breastfeeding | Birth to six months postpartum
  Prevalence of infants exclusively breastfed using maternal reports and the deuterium dose-to-mother technique (in a subgroup)
Dietary intake during six months pregnancy | Assessed at 6 months and 9 months pregnancy
  Prevalence of women with adequate dietary intake during six months pregnancy
Dietary intake at six months post-partum | Assessed at six months postpartum
  Prevalence of women with adequate dietary intake at six months post-partum

SECONDARY OUTCOMES:
Gestational weight gain | Gestational weight gain will be measured in all pregnant women at six and nine months pregnancy
  Weight gain at term (Kg)
Maternal genital infections | Maternal genital infections will be assessed at nine months pregnancy
  The presence of genital infections that are known to affect a healthy pregnancy, including but not limited to bacterial vaginosis, Chlamydia trachomatis, Neisseria gonorrhoeae, Trichomonas vaginalis, Listeria monocytogenes.
Birth weight | Birth weight will be assessed in all newborns
  Birth weight (g)
Infant weight | Weight of infants will be assessed monthly from birth until six months of age
  Infant weight (g) on a monthly basis
Infant length | Length of infants will be assessed monthly from birth until six months of age
  Infant length (cm) on a monthly basis
Infant anemia | Hemoglobin concentrations will be measured at six months of age
  Hemoglobin concentrations (g/dL)
Maternal parasitic infections | Worm infections will be assessed in all women at 6 months pregnancy, 9 months pregnancy, and at two weeks- and 6 months post partum
  The presence of worm parasites and egg density in the stools. Three common parasites and their eggs will be investigated, i.e. Ascaris lumbricoides (round worm), Trichuris trichiura (whipworm) and Ancyclostoma duodenale or Necater americanus (hookworms).
Infant parasitic infections | Infant parasitic infections will be assessed at 6 months of age.
  The prevalence of Giarida and Cryposporidium will be assessed in all infants
Maternal plasma ferritin | Plasma ferritin is assessed in a subgroup of women at 9 months pregnancy and at six months postpartum
  Iron status as indicated plasma ferritin (micro_g/L) is a test to evaluate iron stores
Infant plasma ferritin | Plasma ferritin is assessed in a subgroup of infants at six months of age
  Iron status as indicated plasma ferritin (micro_g/L) is a test to evaluate iron stores
Maternal soluble transferrin receptor | Plasma ferritin is assessed in a subgroup of women at 9 months pregnancy and at six months postpartum
  Soluble transferrin receptor (mg/L) is an indicator for iron deficiency especially in high inflammation settings
Infant soluble transferrin receptor | Soluble transferrin receptor is assessed in a subgroup of infants at six months of age
  Soluble transferrin receptor (mg/L) is an indicator for iron deficiency especially in high inflammation settings
Maternal serum concentrations in Vitamin A (retinol) | Serum concentrations in Vitamin A are assessed in a subgroup of women at 9 months pregnancy and at six months postpartum
  Retinol concentrations in serum is an indicator of vitamin A status
Infant serum concentrations in Vitamin A (retinol) | Serum concentrations in Vitamin A are assessed in a subgroup of infants at six months of age
  Retinol concentrations in serum is an indicator of vitamin A status
Maternal serum concentrations in vitamin B12 | Vitamin B12 concentrations will be assessed in a subgroup of women at 9 months pregnancy and at six months postpartum
  Serum concentrations in vitamin B12
Infant serum concentrations in vitamin B12 | Vitamin B12 concentrations will be assessed in a subgroup of infants at six months of age
  Serum concentrations in vitamin B12

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan De Henauw, Md. PhD, Principal Investigator — University Ghent; Souheila Abbeddou, MSc. PhD, Principal Investigator — University Ghent; Bruno Levecke, PhD, Principal Investigator — University Ghent
Locations (1):
- Arba Minch University, Arba Minch, Dirashe District, Ethiopia

IPD SHARING:
Plan to Share IPD: No
All the data that can affect the main or the secondary outcomes will be used in the analyses and shared as necessary.
  Data on helminthic infection will use household characteristics and women and infants nutritional status

REFERENCES:
- [Background] Lassi ZS, Salam RA, Haider BA, Bhutta ZA. Folic acid supplementation during pregnancy for maternal health and pregnancy outcomes. Cochrane Database Syst Rev. 2013 Mar 28;2013(3):CD006896. doi: 10.1002/14651858.CD006896.pub2. PMID 23543547
- [Background] Rasmussen KM, Stoltzfus RJ. New evidence that iron supplementation during pregnancy improves birth weight: new scientific questions. Am J Clin Nutr. 2003 Oct;78(4):673-4. doi: 10.1093/ajcn/78.4.673. No abstract available. PMID 14522723
- [Background] Brooker S, Bethony J, Hotez PJ. Human hookworm infection in the 21st century. Adv Parasitol. 2004;58:197-288. doi: 10.1016/S0065-308X(04)58004-1. PMID 15603764
- [Background] Prociv P, Luke RA. Evidence for larval hypobiosis in Australian strains of Ancylostoma duodenale. Trans R Soc Trop Med Hyg. 1995 Jul-Aug;89(4):379. doi: 10.1016/0035-9203(95)90016-0. No abstract available. PMID 7570868
- [Background] Asundep NN, Jolly PE, Carson AP, Turpin CA, Zhang K, Wilson NO, Stiles JK, Tameru B. Effect of Malaria and Geohelminth Infection on Birth Outcomes in Kumasi, Ghana. Int J Trop Dis Health. 2014;4(5):582-594. doi: 10.9734/IJTDH/2014/7573. PMID 25414840
- [Background] Kavle JA, Landry M. Addressing barriers to maternal nutrition in low- and middle-income countries: A review of the evidence and programme implications. Matern Child Nutr. 2018 Jan;14(1):e12508. doi: 10.1111/mcn.12508. Epub 2017 Aug 24. PMID 28836343
- [Background] Verstraelen H, Delanghe J, Roelens K, Blot S, Claeys G, Temmerman M. Subclinical iron deficiency is a strong predictor of bacterial vaginosis in early pregnancy. BMC Infect Dis. 2005 Jul 6;5:55. doi: 10.1186/1471-2334-5-55. PMID 16000177
- [Background] Tuddenham S, Ghanem KG, Caulfield LE, Rovner AJ, Robinson C, Shivakoti R, Miller R, Burke A, Murphy C, Ravel J, Brotman RM. Associations between dietary micronutrient intake and molecular-Bacterial Vaginosis. Reprod Health. 2019 Oct 22;16(1):151. doi: 10.1186/s12978-019-0814-6. PMID 31640725
- [Background] Ashorn P, Hallamaa L, Allen LH, Ashorn U, Chandrasiri U, Deitchler M, Doyle R, Harjunmaa U, Jorgensen JM, Kamiza S, Klein N, Maleta K, Nkhoma M, Oaks BM, Poelman B, Rogerson SJ, Stewart CP, Zeilani M, Dewey KG. Co-causation of reduced newborn size by maternal undernutrition, infections, and inflammation. Matern Child Nutr. 2018 Jul;14(3):e12585. doi: 10.1111/mcn.12585. Epub 2018 Jan 8. PMID 29316198
- [Result] Bhutta ZA, Das JK, Rizvi A, Gaffey MF, Walker N, Horton S, Webb P, Lartey A, Black RE; Lancet Nutrition Interventions Review Group, the Maternal and Child Nutrition Study Group. Evidence-based interventions for improvement of maternal and child nutrition: what can be done and at what cost? Lancet. 2013 Aug 3;382(9890):452-477. doi: 10.1016/S0140-6736(13)60996-4. Epub 2013 Jun 6. PMID 23746776
- [Derived] Boynito WG, Worsa KT, Gutema BT, Yeshitila YG, Tessema GY, Yohanis T, Henauw S, Cools P, Levecke B, Abbeddou S. Effects of Video-Based Health Education on Birth Outcomes and Anaemia Status of Mothers in Dirashe District South Ethiopia: A Cluster Randomized Controlled Trial. Matern Child Nutr. 2025 Sep 24:e70122. doi: 10.1111/mcn.70122. Online ahead of print. PMID 40990120
- [Derived] Godana Boynito W, Tessema GY, Temesgen K, De Henauw S, Abbeddou S. Acceptability and feasibility of video-based health education for maternal and infant health in Dirashe District, South Ethiopia: A qualitative study. PLOS Glob Public Health. 2023 Jun 29;3(6):e0000821. doi: 10.1371/journal.pgph.0000821. eCollection 2023. PMID 37384600
- See also: Evidence of Effective Approaches to Social and Behavior Change Communication for Preventing and Reducing Stunting and Anemia: Report from a Systematic Literature Review — https://www.spring-nutrition.org/sites/default/files/publications/series/spring_sbcc_lit_review.pdf